CLINICAL TRIAL: NCT00545441
Title: A Randomized Clinical Trial Comparing Surgisis AFP to Advancement Flap for the Repair of Anal Fistulas
Acronym: Surgisis® AFP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Collaborators: Cook Biotech Incorporated (Industry); Cook Ireland, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-006
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2014-10-29 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Anal Fistula
Keywords: Anal fistula; fistula in ano; anorectal fistula
MeSH Terms: conditions — Rectal Fistula | interventions — Surgical Flaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Surgisis® AFP
  Interventions: Device: Surgisis Biodesign Anal Fistula Plug (Surgisis® AFP)
- 2 (Active Comparator): Flap
  Interventions: Device: Flap

INTERVENTIONS:
Device: Surgisis Biodesign Anal Fistula Plug (Surgisis® AFP) — Surgical placement of the Surgisis AFP is performed under general anesthesia.
  Other Names: Surgisis Biodesign
  Arms: 1
Device: Flap — Advancement flap surgery is performed; no anal fistula plug is placed
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether the Surgisis anal fistula plug is just as effective in healing anal fistulas as compared to the advancement flap procedure.

ELIGIBILITY:
Inclusion Criteria:

* Over eighteen years old
* Clinical diagnosis of primary anal fistula categorized as transsphincteric, suprasphincteric, or extrasphincteric in nature
* Pre-placement of seton required for at least 6 weeks prior to surgical treatment
* Willing to sign informed consent and share data with study sponsor and Surgisis AFP manufacturer

Exclusion Criteria:

* Recurrent fistula tracts
* J-pouch fistulas
* Superficial fistulas
* Fistulas with active abscess, infection, or acute inflammation
* History of Chron's Disease
* History of Ulcerative Colitis
* History of HIV or other immune system disease
* History of collagen disease
* History of radiation to the anorectal region
* Allergies to pig tissue or pig products
* Religious or cultural objection to the use of pig tissue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2008-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Schwandner, MD, Principal Investigator — Justus-Liebig-Universitat Giessen
Locations (6):
- Germany (6):
  - Justus-Liebig-Universitat Giessen, Giessen, Giessen
  - Krankenhaus Waldfriede, Berlin
  - End-und Dickdarmzentrum Hannover, Hanover
  - Enddarmzentrum Mannheim, Mannheim
  - Caritas-Krankenhaus St. Joseph, Regensburg
  - St. Joseph Hospital, Wiesbaden

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgisis® AFP: Surgisis Biodesign Anal Fistula Plug (SurgiSIS AFP): Surgical placement of the Surgisis AFP is performed under general anesthesia.
Period: Overall Study
Arm/Group | Surgisis® AFP | Flap
Started | 44 | 42
Completed | 26 | 26
Not Completed | 18 | 16
Not completed — Fistula draining at 6 months | 2 | 4
Not completed — Lost to Follow-up | 9 | 5
Not completed — Technical failure | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Persistence or recurrence of fistula | 5 | 2
Not completed — Patients were not treated | 1 | 3

BASELINE CHARACTERISTICS:
Population: Patients that were not treated were not included in the analysis. There was 1 patient in the Surgisis arm and 3 patients in the Flap arm that were not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Surgisis® AFP | Flap | Total
Number analyzed (Participants) | 43 | 39 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] — One patient in the SurgiSIS AFP arm has age missing.
  years | 45.1 (13.2) | 49.4 (13.1) | 47.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 33 | 23 | 56

OUTCOME MEASURES:

1. Primary Outcome: Healing Success
Description: Healing was defined as "closure of external opening with absence of abscess, drainage and pain."
Time Frame: 12 months
Population: Patients that were lost to follow-up, withdrew, or not treated were not included in the analysis. In the Surgisis arm, there were 9 patients lost to follow-up, 1 patient withdrew, and 1 patient not treated; in the Flap arm, there were 5 patients lost to follow-up, 1 patient withdrew, and 3 patients not treated.
Measure: Number; unit: participants
Arm/Group | Surgisis® AFP | Flap
Number analyzed (Participants) | 33 | 33
participants | 22 | 25
Statistical Analysis 1: Comparison: Surgisis® AFP vs Flap; Test type: Non-Inferiority or Equivalence — Alpha = 0.05 and power = 0.8, a non-inferiority margin of 10%; p = 0.59, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Surgisis® AFP | Flap
Serious Adverse Events (participants affected / at risk) | 1/43 | 2/39
Other Adverse Events (participants affected / at risk) | 7/43 | 5/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgisis® AFP (N=43) | Flap (N=39)
Induration / Redness / Swelling Involving External Opening (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fistula Tract Re-Opened After Closure had been Documented (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Newly apparent fistula opening (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgisis® AFP (N=43) | Flap (N=39)
Fistula tract re-opened after closure had been documented (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Induration / Redness / Swelling involving external opening (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Infection / Abscess involving fistula (Infections and infestations) | 3 (3) | 3 (5)
Plug fell out or flap failed (Surgical and medical procedures) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days